CLINICAL TRIAL: NCT04252404
Title: FranceLEVO - Zimino® Registry: a French Registry Evaluating the Use of Levosimendan (Zimino®)
Brief Title: FranceLEVO - Zimino Registry (FZR)
Acronym: FZR
Status: Completed | Type: Observational
Sponsor: Arcothova (Other)
Responsible Party: Principal Investigator, Cholley Bernard, Coordinating Investigator, Arcothova
Other Study IDs: Arcothova
Record Dates: First submitted 2020-01-15; First posted 2020-02-05 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Acute Heart Failure
Keywords: low cardiac output syndrome; cardiogenic shock
MeSH Terms: conditions — Cardiac Output, Low; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The French National Authority for Health (Haute Autorité de santé) requested a registry study to obtain post-market surveillance data to describe baseline clinical profiles, management and outcome of patients treated with Zimino®. This study is designed to provide real-life data on the use, safety and clinical outcomes of Zimino® in routine clinical practice in France.

DETAILED DESCRIPTION:
This is a real-life, non-interventional, observational, multicentre study in all patients (including children) receiving Zimino® in France.

The patients will be evaluated during the index hospitalisation and on follow-up days 30 (±15) and 90 (±15) after hospital discharge. The follow-up can be a phone call or a visit to the hospital. Patients who meet the eligibility criteria will be identified consecutively at each hospital. The participating hospitals will vary in size and medical activities, depending on their location and the population size they serve.

The physician will determine the patient's treatment strategy. Drug prescriptions and the indications to perform diagnostic or therapeutic procedures will be left completely to the discretion of the physicians.

The estimated enrollment period is 12 months (enrollment of the first patient - enrollment of the last patient), or less if the cohort (n=600) is completed earlier, and the maximum total data collection period is 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving Zimino® treatment
* Patients or patient's families not objecting to the patient's participation in the study.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cardiac dysfunction receiving levosimendan (Zimino®)
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Indication for levosimendan (Zimino) | from January 28, 2020 until January 28, 2021
  Physicians will be requested to choose one of the following indications (pop-up list):
  1. Cardiogenic shock (medical setting or post cardiac surgery)
  2. Heart failure decompensation (medical, setting)
  3. Low cardiac output syndrome (post cardiac surgery)
  4. Heart failure decompensation in a patient receiving beta-blockers
  5. ECMO weaning
  6. Repetitive use in a patient with end-stage heart failure
  7. Other (text)
Dose of levosimendan (Zimino) (in µg/kg/min) | from January 28, 2020 until January 28, 2021
  Physicians will be requested to describe the levosimendan regimen used:
  A) Loading dose (in µg/kg) B) Dose of the continuous infusion (in µg/kg/min)
Duration of levosimendan (Zimino) infusion | from January 28, 2020 until January 28, 2021
  Number of hours during which the patient received levosimendan

CONTACTS AND LOCATIONS:
Overall Officials: Bernard CHOLLEY, MD, PhD, Principal Investigator — Arcothova
Locations (1):
- Hôpital Européen Georges Pompidou, AP-HP, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No
The data will remain with the sponsor (Arcothova)

DOCUMENTS (2):
  • Study Protocol (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT04252404/Prot_000.pdf
  • Informed Consent Form (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT04252404/ICF_001.pdf